CLINICAL TRIAL: NCT02681367
Title: The First Study to Compare the Effect of Freeze All Policy Versus Fresh Embryo Transfer After ICSI in Patients With Recurrent Implantation Failure
Brief Title: Management of Recurrent Implantation Failure
Acronym: RIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TopLab Company for ART Laboratories Consultation and Training (Other)
Responsible Party: Principal Investigator, Yasmin Magdi, Research and development department director, TopLab Company for ART Laboratories Consultation and Training
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #001008
Record Dates: First submitted 2016-02-08; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Recurrent Implantation Failure (RIF)
Keywords: Recurrent implantation failure; Freeze all policy; endometrial receptivity; implantation; clinical outcome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fresh embryo transfer (No Intervention): Patient with RIF underwent ICSI cycle followed by Day 5 fresh embryo transfer.
- Freeze all (Experimental): Patient with RIF. All of them underwent ICSI cycle, all their embryos were cryopreserved at Day 5 and transferred in a consecutive natural cycle.
  Interventions: Other: Freeze all policy

INTERVENTIONS:
Other: Freeze all policy — Cryopreservation of human blastocysts for freeze all group has been employed using vitrification. The blastocysts were transferred after thawing in a frozen-thawed cycle.
  Other Names: Frozen-thawed embryo transfer
  Arms: Freeze all

SUMMARY:
This is the first study to investigate, whether pregnancy and implantation rates would improve in patients with recurrent implantation failure (RIF), if all embryos were to be frozen and transferred in a consecutive natural cycle.

DETAILED DESCRIPTION:
There is growing evidence that elective frozen-thawed embryo transfer in a non-stimulated cycle (freeze-all policy) would eliminate the risk of controlled ovarian stimulation and resulting in better endometrial receptivity and lower uterine contractility as compared with fresh intracytoplasmic sperm injection (ICSI) cycles.

RIF refers to women who fail to achieve a clinical pregnancy, in a minimum of three embryo transfer cycles with at least four good-quality embryos were transferred in a woman < 40 years. It affects approximately 10% of ICSI cases. Many management protocols aimed to enhance ICSI outcome in cases of RIF, however, none of them examined the effect of freeze all policy in this category of patients.

ELIGIBILITY:
Inclusion Criteria:

1. gonadotropin-releasing hormone agonist and recombinant follicle-stimulating hormone (FSH) in a long protocol cycles;
2. female partners were under age of 40 years;
3. all the patients had a history of recurrent implantation failure i.e: failed to achieve a clinical pregnancy after at least three fresh ICSI cycles where at least 8 good embryos were transferred;
4. their embryos were pushed to Day 5 resulting in blastocysts, and undergo embryo transfer day 5 or vitrification on day 5;
5. endometrial thickness ≥ 7 mm;
6. selected embryos for embryo transfer were blastocysts. -

Exclusion Criteria:

Couples with testicular or epididymal sperm were excluded.

-

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks post embryo transfer
  Clinical pregnancy was identified by fetal cardiac activity on ultrasound examination 4 weeks after embryo transfer.

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 10 weeks post embryo transfer
  Ongoing pregnancy rate was defined as the number of pregnancies with visible fetal heart motion over the number of transferred embryos at 10 weeks' gestation.
Implantation rate | 6 weeks after embryo transfer
  Implantation rate was defined as the number of intrauterine gestational sacs over the total number of embryos transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Magdi, M.Sc, Principal Investigator — Research and development department director at TopLab Company for ART laboratories consultations and training

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Timeva T, Shterev A, Kyurkchiev S. Recurrent implantation failure: the role of the endometrium. J Reprod Infertil. 2014 Oct;15(4):173-83. PMID 25473625
- [Result] Roque M. Freeze-all policy: is it time for that? J Assist Reprod Genet. 2015 Feb;32(2):171-6. doi: 10.1007/s10815-014-0391-0. Epub 2014 Nov 27. PMID 25428436
- [Result] Simon A, Laufer N. Assessment and treatment of repeated implantation failure (RIF). J Assist Reprod Genet. 2012 Nov;29(11):1227-39. doi: 10.1007/s10815-012-9861-4. Epub 2012 Sep 14. PMID 22976427